CLINICAL TRIAL: NCT04565366
Title: Early Critical Care Decisions and Outcomes After SCI: TRACK-SCI
Brief Title: Transforming Research and Clinical Knowledge in Spinal Cord Injury
Acronym: TRACK-SCI
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); The Craig H. Neilsen Foundation (Other); Wings for Life (Other)
Responsible Party: Sponsor
Other Study IDs: SC150198; W81XWH-16-1-0497 (Other Grant/Funding Number: United States Department of Defense)
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injury; Biomarkers; Neuroimaging; NINDS Common Data Elements; Spine Injury; Neurosurgery; Neurology
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, CSF, and white blood cells (WBCs) will be collected at the time closest to injury, Day 2, Day 3, and Day 5 if patient is in the hospital. Serum and WBCs will be collected at 6 months and 12 months post-injury. Samples will be banked at -80 degrees Celsius.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Spinal Cord Injury: Individuals recently admitted to hospital and diagnosed with acute, traumatic spinal cord injury.
- Trauma Control: Individuals recently admitted to hospital and diagnosed with an acute, traumatic injury that is not spinal cord injury.
- Healthy Control: Generally healthy individuals not recently diagnosed with an acute, traumatic injury (including spinal cord injury).

SUMMARY:
The overall goal of Transforming Research and Clinical Knowledge in Spinal Cord Injury (TRACK-SCI) study is to determine the relationships among the clinical, neuroimaging, cognitive, genetic and proteomic biomarker characteristics of acute traumatic spinal cord injury (SCI). TRACK-SCI seeks to combine high quality care variables with high density physiology data collection to better understand diagnose, characterize, and track the temporal profile of recovery for SCI patients. The Investigators are enrolling patients within 24 hours of injury who present to a TRACK-SCI site with a spinal cord injury that meets eligibility criteria.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is a major cause of morbidity worldwide with debilitating impacts on quality of life and the healthcare system. To date, a data-dense research registry specific to SCI remains to be constructed. To this end, the study will collect SCI data across five primary domains: 1) demographics and baseline history, 2) clinical course variables from the emergency department (ED) to the intensive care unit (ICU), 3) standard of care neuroimaging (CT and MRI) and intraoperative neuromonitoring, 4) blood and cerebrospinal fluid (CSF) samples for proteomic and genetic biomarkers, and 5) outcome measures of functional disability, mental health and quality of life at 3, 6, and 12 months. The investigators seek to correlate these high-density physiology data with baseline risk factors, imaging parameters, and biomarkers for a comprehensive approach to SCI diagnosis during acute care as well as prognosis across subacute and chronic phases of recovery -- in order to truly step toward the advancement of research and clinical knowledge in SCI.

The main objective is to provide a comprehensive prospective analysis of multiple variables in acute SCI that impact long-term outcomes. This is intended to provide a rich resource for asking key questions related to the optimization of treatment, and the planning and execution of pivotal clinical trials in SCI.

Core Hypotheses:

1. Multiple critical care variables will be predictive of both sensorimotor and autonomic outcomes, and susceptibility to infections at discharge and 6 and 12 mos after injury.
2. Quantitative MRI indices of cord damage, and biomarkers of acute immune responses to injury will predict neurological outcomes at discharge and at 6 and 12 mos.
3. The multivariate analysis of the constellation of acute variables and long-term outcome measures will yield new derived predictors of outcome that will facilitate stratification for clinical trials.

Specific Aims:

Aim 1. Diagnosis: Building a knowledge network for acute SCI. A detailed prospective study of critical care practices and outcomes for SCI patients admitted to TRACK-SCI sites will be conducted to build a knowledge network for acute SCI diagnostics.

Aim 2. Prognosis: Predictive models and biomarkers. The research team will develop multidimensional prognostic indicators for predicting outcomes and stratifying patients using detailed physiological, imaging, and genetic datasets.

Aim 3: Data analysis and sharing. The development of better predictors of outcome and methods for stratification will be advanced by allowing qualified access to our granular data. The availability to qualified users of the detailed acute 'diagnostic' dataset along with gene-expression data and functional outcomes at 6&12 mos will leverage the project as a valuable international SCI community resource.

ELIGIBILITY:
Inclusion Criteria:

* For SCI group: individuals at least 18 years of age recently diagnosed with acute, traumatic spinal cord injury
* For Trauma Control group: individuals at least 18 years of age recently diagnosed with acute, traumatic injury that is not spinal cord injury
* For Healthy Control group: generally healthy individuals at least 18 years of age not recently diagnosed with acute, traumatic injury (including SCI)

Exclusion Criteria:

* Individuals who are pregnant
* Individuals who are in-custody/prisoners
* Individuals who are under psychiatric hold
* For non-SCI individuals, they must not have had a spinal cord injury in the past
* For non-SCI individuals, they must not have a history of previous central nervous system injury (i.e. stroke, spinal cord injury, traumatic brain injury, seizures, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will enroll patients presenting to the Emergency Department with an acute SCI, in which the patient has sustained a traumatically induced disruption of spinal cord function, as manifested by one of the following: detection through clinical assessment of motor and/or sensory deficit from baseline, and/or radiologic evidence of cord signal disruption.
  For trauma controls, investigators will recruit non-neurological traumatic injury patients from the ED. For healthy controls, investigators will recruit primarily friends and family members of SCI participants.
Sampling Method: Non-Probability Sample
Enrollment: 726 (Estimated)
Dates: Start 2015-05-14 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Gene expression level in number of messenger RiboNucleic Acid (mRNA) transcripts for all genes expressed in white blood cells | Baseline (healthy control group), or as close as possible to time of injury (SCI and trauma control group)
  Obtained from a 4.0mL blood draw
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) (SCI Only) | From admission to 12 months post-injury
  American Spinal Injury Association standard assessment for documentation of the level and severity of a spinal cord injury (SCI). The ISNCSCI yields a grade from A to D, wherein A indicates greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Beattie, PhD, Principal Investigator — University of California, San Francisco
Locations (5):
- United States (5):
  - University of California, San Francisco - Fresno, Fresno, California
  - University of California, San Francisco, San Francisco, California
  - Ohio State University, Columbus, Ohio
  - University of Utah, Salt Lake City, Utah
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
All data (de-identified) that underlie results in a publication will be made available to other researchers upon Executive Committee approval. Select de-identified datasets will be made publicly available via the Open Data Commons for Spinal Cord Injury (ODC-SCI), accessible at <https://scicrunch.org/odc-sci>.
Time Frame: Eligible datasets will become available starting 6 months after publication.
Access Criteria: Select de-identified datasets will be made available to qualified researchers upon review and approval of a Data Collaboration Request by the TRACK-SCI Executive Committee. Eligible publicly accessible de-identified datasets will be available through ODC-SCI.

REFERENCES:
- [Background] Talbott JF, Whetstone WD, Readdy WJ, Ferguson AR, Bresnahan JC, Saigal R, Hawryluk GW, Beattie MS, Mabray MC, Pan JZ, Manley GT, Dhall SS. The Brain and Spinal Injury Center score: a novel, simple, and reproducible method for assessing the severity of acute cervical spinal cord injury with axial T2-weighted MRI findings. J Neurosurg Spine. 2015 Oct;23(4):495-504. doi: 10.3171/2015.1.SPINE141033. Epub 2015 Jul 10. PMID 26161519
- [Background] Burke JF, Yue JK, Ngwenya LB, Winkler EA, Talbott JF, Pan JZ, Ferguson AR, Beattie MS, Bresnahan JC, Haefeli J, Whetstone WD, Suen CG, Huang MC, Manley GT, Tarapore PE, Dhall SS. Ultra-Early (<12 Hours) Surgery Correlates With Higher Rate of American Spinal Injury Association Impairment Scale Conversion After Cervical Spinal Cord Injury. Neurosurgery. 2019 Aug 1;85(2):199-203. doi: 10.1093/neuros/nyy537. PMID 30496474
- [Background] Tsolinas RE, Burke JF, DiGiorgio AM, Thomas LH, Duong-Fernandez X, Harris MH, Yue JK, Winkler EA, Suen CG, Pascual LU, Ferguson AR, Huie JR, Pan JZ, Hemmerle DD, Singh V, Torres-Espin A, Omondi C, Kyritsis N, Haefeli J, Weinstein PR, de Almeida Neto CA, Kuo YH, Taggard D, Talbott JF, Whetstone WD, Manley GT, Bresnahan JC, Beattie MS, Dhall SS. Transforming Research and Clinical Knowledge in Spinal Cord Injury (TRACK-SCI): an overview of initial enrollment and demographics. Neurosurg Focus. 2020 May 1;48(5):E6. doi: 10.3171/2020.2.FOCUS191030. PMID 32357323
- [Background] Dhall SS, Haefeli J, Talbott JF, Ferguson AR, Readdy WJ, Bresnahan JC, Beattie MS, Pan JZ, Manley GT, Whetstone WD. Motor Evoked Potentials Correlate With Magnetic Resonance Imaging and Early Recovery After Acute Spinal Cord Injury. Neurosurgery. 2018 Jun 1;82(6):870-876. doi: 10.1093/neuros/nyx320. PMID 28973360
- [Background] McCoy DB, Dupont SM, Gros C, Cohen-Adad J, Huie RJ, Ferguson A, Duong-Fernandez X, Thomas LH, Singh V, Narvid J, Pascual L, Kyritsis N, Beattie MS, Bresnahan JC, Dhall S, Whetstone W, Talbott JF; TRACK-SCI Investigators. Convolutional Neural Network-Based Automated Segmentation of the Spinal Cord and Contusion Injury: Deep Learning Biomarker Correlates of Motor Impairment in Acute Spinal Cord Injury. AJNR Am J Neuroradiol. 2019 Apr;40(4):737-744. doi: 10.3174/ajnr.A6020. Epub 2019 Mar 28. PMID 30923086